CLINICAL TRIAL: NCT02965911
Title: A Randomized Controlled Clinical Trial on the Efficacy and Safety of Fenofibrate Combined With Ursodeoxycholic Acid in PBC Patients With an Incomplete Biochemical Response to UDCA
Brief Title: Efficacy and Safety of Fenofibrate Combined With UDCA in PBC Patients With an Incomplete Biochemical Response to UDCA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJ302-FGRXGB-002
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Primary Biliary Cirrhosis
Keywords: UDCA, Fenofibrate
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UDCA Standard treatment (Active Comparator): All subjects will reiceive UDCA at a dose of 13-15mg/kg/d by oral for 12 months, and UDCA will be maintained after 12 months.
  Interventions: Drug: UDCA
- Fenofibrate Combined with UDCA Treatment (Experimental): All subjects will be treated with UDCA,13-15mg/kg/d, and Fenofibrate, 200mg/d by oral for 12 month,
  Interventions: Drug: Fenofibrate; Drug: UDCA

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate is a drug of the fibrate class. it reduces both low-density lipoprotein (LDL) and very low density lipoprotein (VLDL) levels, as well as increasing high-density lipoprotein (HDL) levels and reducing triglyceride levels.
  Other Names: Antara, Fenoglide, Fibricor, Lipofen, Lofibra
  Arms: Fenofibrate Combined with UDCA Treatment
Drug: UDCA — Ursodeoxycholic acid，the abbreviation UDCA, is one of the secondary bile acids, which are metabolic byproducts of intestinal bacteria，it is the only FDA approved drug to treat PBC.
  Other Names: Ursa，Urso, Urso Forte, Ursocol, Ursofalk,

SUMMARY:
The purpose of this protocol is to conduct a trial in a selected population of patients with PBC based on an incomplete biochemical response after 12 months of UDCA therapy.

DETAILED DESCRIPTION:
Primary biliary cholangitis is a chronic cholestatic liver disease, ursodeoxycholic acid (UDCA) is the only drug approved for the treatment of PBC. Although UDCA can improve the clinical outcomes in patients with PBC, about 40% of PBC patients show an incomplete biochemical response to this treatment, accordingly have a significantly increased risk of developing liver transplantation or death. Therefor there is a urgently needed for better therapies for these patients. The development of new treatments is therefore needed. The Fenofibrate is the candidate, there is now a substantial body of circumstantial evidence supporting that Fenofibrate is well tolerated and can improve biochemical response in PBC patients with incompleted response to UDCA. The purpose of this protocol is to conduct a trial in a selected population of patients with PBC based on an incomplete biochemical response after 12 months of UDCA therapy.

ELIGIBILITY:
Inclusion Criteria:

1. PBC Patient , previous treatment with UDCA 13-15 mg/kg/day for at least 1 year, showed incomplete biochemical response;
2. Patients who showing an incomplete biochemical response to UDCA as defined by: ALP > 3ULN,AST> 2N ,total bilirubin >17 µmol/l after ≥ 12 months of UDCA at the dose of 13 - 15 mg/kg/day.

3,signed informed consent after careful review of information and study details.

Exclusion Criteria:

1. Hypersensitivity to fenofibrate
2. Administration of the following drugs at any time during the 3 months prior to screening for the study: methotrexate, colchicines, azathioprine, systemic steroids.
3. Decompensation PBC, such as recurrent variceal hemorrhage, uncontrolled encephalopathy or refractory ascites
4. Anticipated need for liver transplantation within one year
5. Co-existing liver diseases such as acute or chronic viral hepatitis, alcoholic liver disease, choledocholithiasis, autoimmune hepatitis, biopsy-proven non-alcoholic fatty liver disease, Wilson's disease and hemochromatosis
6. Acute or chronic renal failure
7. Known history of cholecystitis with intact gallbladder
8. Pregnant or nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2021-09-08 (Estimated); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Serum Level of Alkaline Phosphatase(ALP) value | 12 months
  To analyze the clinical efficacy of UDCA combined with UDCA at 1 year compared to baseline values.

SECONDARY OUTCOMES:
Total bilirubin(TBIL) value | 12 months
  To analyze the clinical efficacy of UDCA combined with UDCA at 1 year compared to baseline values.
Aspartate aminotransferase(AST) value | 12 months
  To analyze the clinical efficacy of UDCA combined with UDCA at 1 year compared to baseline values.
Serum Level of Gamma-glutamyl transpeptidase (GGT) value | 12 months
  To analyze the clinical efficacy of UDCA combined with UDCA at 1 year compared to baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengsheng Zou, Dr., Study Director — Beijing 302 Hospital
Locations (1):
- Beijing 302 hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No